CLINICAL TRIAL: NCT06004063
Title: Safety, Tolerability, and Efficacy of Enteral Nutrition Versus Standard of Care Nutrition in Hematopoietic Stem Cell Transplant Patients: A Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-0116; NCI-2023-06448 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Stem Cell
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral nutrition (EN)-Group 1 (Experimental): Participants will receive enteral feeding (directly into the stomach) based on your ability to receive your daily caloric needs by mouth. Participants will be monitored by a dietician and may receive feeding by vein to achieve caloric goals.
  Interventions: Dietary Supplement: Enteral nutrition (EN); Other: Standard care parenteral nutrition (PN)
- Standard care parenteral nutrition (PN)-Group 2 (Active Comparator): Participants will receive the standard of care. Participants will be monitored by a dietician to see if the participants are able to receive your daily caloric needs by mouth. Some participants may be able to receive oral dietary supplements, but if this is not possible or not enough, participants will begin receiving standard of care feeding by vein.
  Interventions: Other: Standard care parenteral nutrition (PN)

INTERVENTIONS:
Dietary Supplement: Enteral nutrition (EN) — Given by Nasogastric Tube
  Arms: Enteral nutrition (EN)-Group 1
Other: Standard care parenteral nutrition (PN) — Given by PO or Given by IV (vein)

SUMMARY:
The goal of this research study is to learn if feeding someone after a stem cell transplant is safe and practical.

DETAILED DESCRIPTION:
Primary Objective:

a. To determine the feasibility, acceptability, and safety of NG tube feeding compared with patients not electing NG tube feeding.

Secondary Objectives:

1. Determine the differential effects of enteral feeding versus Parenteral feeding on nutrition, and quality of life.
2. Determine the differential effects of enteral feeding versus parenteral feeding on survival and, medical comorbidities
3. Determine the differential effects of enteral feeding versus parenteral feeding on Fitbit data study for patients co-enrolled in Pediatric Energy Balance Data Repository Protocol PA18-0130.
4. Identify differential effects on microbiome for patients co-enrolled on MDACC protocol 2014-0938 "Longitudinal Biospecimen Acquisition for All Tumor Types And At-Risk Tissue
5. Determine adverse effects of enteral feeding in this population

ELIGIBILITY:
Inclusion Criteria:

1. Have plans to be admitted or be admitted to an inpatient pediatric or adult ward for the purpose of HSCT.
2. Be greater than 2 years of age and less than 25 years of age at time of study enrollment.
3. Participants > 18 or guardians for participants < 18 are willing and able to give written informed consent and to comply with all of the study activities. Assent is required for children > 7 years old.

   a) Participants must be English, Italian, Chinese/Mandarin, or Spanish speaking
4. Participants will be encouraged to co-enroll on two additional related energy -balance protocols (highly encouraged but not required)

   1. MDACC protocol PA18-0130. This protocol will enable us to track physical activity through their receipt of a Fitbit (Pediatric Energy Balance Data Repository Protocol.) , and
   2. MDACC protocol LAB99-062 "A Study to Collect Peripheral Blood, Tissue, and Bone Marrow samples from Donors and Recipients of blood and marrow transplants for Laboratory Research" which will allow collection of stool for exploration of the effects of feeding on microbiome data specifically.
5. Participants will be asked to consider co-enrollment on Stem Cell Registry study (not required):

   1. PA19-0756: This is a prospective multi-center study to understand the contribution of vascular endothelial dysfunction towards morbidity and mortality among children and adolescents/young adults (AYA) undergoing HCT/CT.

Exclusion Criteria:

1. Patients in whom EN is contraindicated (e.g intestinal ischemia, complete bowel obstruction, or other anatomical obstructive process), or all available routes of EN are contraindicated. Surgical GT placements for the sole purpose of study participation will not be entertained. See Table 1
2. Females who are pregnant. We follow FACT guidelines. Per Foundation for the Accreditation of Cellular Therapy (FACT), female patients must have a negative pregnancy test 7 days prior to bone marrow transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Shehla Razvi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org